CLINICAL TRIAL: NCT02427451
Title: Obinutuzumab, Ibrutinib, and Venetoclax for Relapsed and Previously Untreated Chronic Lymphocytic Leukemia (CLL)
Brief Title: Bcl-2 Inhibitor GDC-0199 in Combination With Obinutuzumab and Ibrutinib in Treating Patients With Relapsed, Refractory, or Previously Untreated Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kerry Rogers (Other)
Responsible Party: Sponsor-Investigator, Kerry Rogers, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-14266; NCI-2015-00252 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-03-04; First posted 2015-04-28 (Estimated); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — venetoclax; obinutuzumab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (obinutuzumab, ibrutinib, Bcl-2 inhibitor GDC-0199) (Experimental): Patients receive obinutuzumab IV on day 1 (days 1, 2, 8, and 15 for course 1 only) every 28 days for up to 8 courses. Beginning in course 2, patients receive ibrutinib PO QD on days 1-28. Beginning in course 3, patients receive Bcl-2 inhibitor GDC-0199 PO QD on days 1-28. Treatment repeats every 28 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bcl-2 Inhibitor GDC-0199; Biological: Obinutuzumab; Drug: Ibrutinib; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Bcl-2 Inhibitor GDC-0199 — Given PO
  Other Names: ABT-0199; ABT-199; GDC-0199; RG7601
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA101; Gazyva; R7159; RO 5072759
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase Ib/II trial studies the best dose and safety of Bcl-2 inhibitor GDC-0199 in combination with obinutuzumab and ibrutinib and to see how well they work in treating patients with chronic lymphocytic leukemia that has returned (relapsed), does not respond to treatment (refractory), or is previously untreated. Bcl-2 inhibitor GDC-0199 and ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as obinutuzumab, may block cancer growth in different ways by targeting certain cells. Giving Bcl-2 inhibitor GDC-0199 together with obinutuzumab and ibrutinib may be a better treatment for chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the dose of venetoclax (Bcl-2 inhibitor GDC-0199) that can be safely administered in combination with obinutuzumab and ibrutinib for the treatment of relapsed/refractory or previously untreated chronic lymphocytic leukemia (CLL).

II. To evaluate the feasibility, safety, and tolerability of venetoclax in combination with obinutuzumab and ibrutinib in patients with relapsed/refractory or previously untreated CLL.

III. To determine the minimal residual disease (MRD)-negative complete response (CR) rate after 12 cycles of treatment with venetoclax in combination with obinutuzumab and ibrutinib in patients with relapsed/refractory or previously untreated CLL.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (ORR) and complete response rate (CR) of venetoclax in combination with obinutuzumab and ibrutinib in patients with relapsed/refractory or previously untreated patients with CLL.

II. To estimate progression free survival (PFS) after treatment with venetoclax in combination with obinutuzumab and ibrutinib in patients with relapsed/refractory or previously untreated patients with CLL.

III. To conduct pharmacokinetic and pharmacodynamic studies of venetoclax in combination with obinutuzumab and ibrutinib in patients with relapsed/refractory or previously untreated patients with CLL.

IV. To examine pre-treatment and serial biomarkers associated with response and mechanisms of resistance to venetoclax, obinutuzumab and ibrutinib when given in combination for relapsed/refractory or previously untreated patients with CLL.

OUTLINE: This is a phase Ib, dose-escalation study of Bcl-2 inhibitor GDC-0199 followed by a phase II study.

Patients receive obinutuzumab intravenously (IV) on day 1 (days 1, 2, 8, and 15 for course 1 only) every 28 days for up to 8 courses. Beginning in course 2, patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Beginning in course 3, patients receive Bcl-2 inhibitor GDC-0199 PO QD on days 1-28. Treatment repeats every 28 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 and 8 weeks, every 3 months for 2 years, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL meeting criteria established in the World Health Organization (WHO) classification of hematologic disorders
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Relapsed or refractory CLL patients must meet the following requirements:

  * Received at least 1 prior therapy
  * Require treatment in the opinion of the investigator
  * Relapsed patients must have developed progressive disease following a response to a prior therapy
  * Refractory patients must have failed to respond or relapsed within 6 months to the last prior therapy
* Treatment-naïve CLL patients must meet the following requirements (Phase II only):

  * Symptomatic disease as defined by International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria
  * Received no prior chemotherapy, immunotherapy, or targeted therapy for the treatment of CLL with the exceptions of palliative loco-regional radiotherapy and corticosteroids for symptom control
* Hemoglobin >= 8 g/dL
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelets >= 40,000/mm^3
* Prothrombin time (PT)/partial thromboplastin time (PTT) =< 1.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN (excepting Gilbert's syndrome)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 × ULN
* Serum creatinine < 2.0 mg/dL or creatinine clearance (Cockcroft) >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Female patients must be surgically sterile, post-menopausal (for at least 1 year), or have negative results from a pregnancy test performed as follows:

  * At screening, on a serum sample obtained within 14 days prior to the first study drug administration, and
  * Prior to dosing, on a urine sample obtained on day 1 of treatment if it has been > 7 days since obtaining the serum pregnancy test result
* All female patients not surgically sterile or post-menopausal (for at least 1 year) and non-vasectomized male patients must practice at least one of the following methods of birth control:

  * Total abstinence from sexual intercourse (minimum one complete menstrual cycle)
  * A vasectomized partner
  * Hormonal contraceptives for at least 2 months prior to day 1 of treatment
  * Double-barrier method
* Non-vasectomized male patients must practice at least one of the following methods of birth control throughout the duration of study participation and for at least 3 months after study treatment:

  * A partner who is surgically sterile or postmenopausal (for at least 1 year) or who is taking hormonal contraceptives (oral, parenteral, vaginal ring, or transdermal) for at least 3 months prior to study drug administration
  * Total abstinence from sexual intercourse
  * Double-barrier method (condom, diaphragm or cervical cup with spermicidal, contraceptive sponge, jellies, or cream)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, immunotherapy, radiotherapy, or investigational therapy within 28 days prior to entering the study or those who have not recovered from adverse events due to agents administered more than 28 days earlier; steroids for control of disease related symptoms are permitted
* Patients who are receiving any other investigational agents
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* Active Richter's transformation
* Known active involvement of the central nervous system by lymphoma or leukemia
* Patients who require warfarin anticoagulation or who have received warfarin or equivalent vitamin K antagonists =< 7 days prior to treatment day 1; patients may be eligible if able to be taken off warfarin and started on an alternative anticoagulant
* Received potent cytochrome P450 3A4 (CYP3A4) inhibitors (such as fluconazole, ketoconazole, and clarithromycin) within 7 days prior to the first dose of study treatment
* Received potent CYP3A4 inducers (such as rifampin, carbamazepine, phenytoin, St. John's wort) within 7 days prior to the first dose of study treatment
* Consumed grapefruit or grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of study treatment
* History of a prior significant toxicity, other than thrombocytopenia, from another Bcl-2 family protein inhibitor
* Known cysteine-481 Bruton's tyrosine kinase (BTK) mutation or CLL refractory to or progressed during ibrutinib or other Cys-481 binding BTK inhibitor treatment
* Known infection with the human immunodeficiency virus (HIV) virus
* A cardiovascular disability status of New York Heart Association class >= 2, defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or angina pain
* Positive hepatitis serology:

  * Hepatitis B virus (HBV): patients with positive serology for hepatitis B defined as positivity for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (anti-HBc); patients who are positive for anti-HBc may be considered for inclusion in the study on a case-by-case basis if they are hepatitis B viral deoxyribonucleic acid (DNA) negative and are willing to undergo ongoing HBV DNA testing by real-time polymerase chain reaction (PCR); patients with positive serology may be referred to a hepatologist or gastroenterologist for appropriate monitoring and management

    * Patients with positive HBSAg consistent with prior vaccination to HBV (i.e., anti-HBs+, anti-HBc-) may participate
    * Patients suspected to have false positive serologic studies because of IV immunoglobulin administration are potentially eligible after negative PCR studies for viral DNA/ribonucleic acid (RNA) and discussion with the principal investigator
  * Hepatitis C (HCV): patients with positive hepatitis C serology unless HCV RNA is confirmed negative and may be considered for inclusion in the study on a case-by-case basis (e.g., patients with negative viral load after HCV-specific treatment)
* History of severe (defined as grade 4 and/or requiring permanent discontinuation of prior antibody therapy) allergic or anaphylactic reactions to human, humanized, chimeric, or murine monoclonal antibodies
* Patients who received a live viral vaccination within 6 months prior to the first dose of study drug
* A female patient who is pregnant or breast-feeding
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of other active malignancies other than CLL within the past 3 years prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma or the cervix uteri or breast
  * Basal cell or localized squamous cell carcinoma of the skin
  * Previous malignancy confirmed and surgically resected (or treated with other modalities) with curative intent or without relapse for >= 2 years
* Vaccination with a live vaccine < 28 days prior to the start of treatment
* Inability to swallow capsules or tablets, or disease significantly affecting gastrointestinal function and/or inhibiting small intestine absorption (malabsorption syndrome, resection of the small bowel, poorly controlled inflammatory bowel disease, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-08-03 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2026-04-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Rogers, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arrato NA, Valentine TR, Byrd JC, Jones JA, Maddocks KJ, Woyach JA, Andersen BL. Illness representations and psychological outcomes in chronic lymphocytic leukaemia. Br J Health Psychol. 2022 May;27(2):553-570. doi: 10.1111/bjhp.12562. Epub 2021 Oct 4. PMID 34608724
- [Derived] Rogers KA, Huang Y, Ruppert AS, Abruzzo LV, Andersen BL, Awan FT, Bhat SA, Dean A, Lucas M, Banks C, Grantier C, Heerema NA, Lozanski G, Maddocks KJ, Valentine TR, Weiss DM, Jones JA, Woyach JA, Byrd JC. Phase II Study of Combination Obinutuzumab, Ibrutinib, and Venetoclax in Treatment-Naive and Relapsed or Refractory Chronic Lymphocytic Leukemia. J Clin Oncol. 2020 Nov 1;38(31):3626-3637. doi: 10.1200/JCO.20.00491. Epub 2020 Aug 14. PMID 32795224
- [Derived] Rogers KA, Huang Y, Ruppert AS, Awan FT, Heerema NA, Hoffman C, Lozanski G, Maddocks KJ, Moran ME, Reid MA, Lucas M, Woyach JA, Whitlow WT, Jones JA, Byrd JC. Phase 1b study of obinutuzumab, ibrutinib, and venetoclax in relapsed and refractory chronic lymphocytic leukemia. Blood. 2018 Oct 11;132(15):1568-1572. doi: 10.1182/blood-2018-05-853564. Epub 2018 Aug 15. PMID 30111609
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients in the phase 1b dose escalation cohorts were enrolled and sequentially assigned to the appropriate dosing cohort. Enrollment was staggered to allow patients to start the ramp up period of venetoclax for the next cohort prior to the completion of the dose-limiting toxicity (DLT) observation period for the previous cohort. However, no patients escalated to a higher target dose until all patients had completed the DLT observation period from the previous cohort.
Groups:
- Phase 1b Cohort 100mg Venetoclax (GDC-0199): Patients receive obinutuzumab IV on day 1 (days 1, 2, 8, and 15 for course 1 only) every 28 days for up to 8 courses. Beginning in course 2, patients receive ibrutinib PO QD on days 1-28. Beginning in course 3, patients receive Bcl-2 inhibitor GDC-0199 PO QD on days 1-28. GDC-0199 is administered through a dose ramp-up throughout course 3 with 20 mg administered in week 1, 50mg in week 2 and 100mg in week 3. The 100mg dose level continues through the rest of the treatment period. Treatment repeats every 28 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.
  Bcl-2 Inhibitor GDC-0199: Given PO
  Obinutuzumab: Given IV
  Ibrutinib: Given PO
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
- Phase 1b Cohort 200mg Venetoclax (GDC-0199): Patients receive obinutuzumab IV on day 1 (days 1, 2, 8, and 15 for course 1 only) every 28 days for up to 8 courses. Beginning in course 2, patients receive ibrutinib PO QD on days 1-28. Beginning in course 3, patients receive Bcl-2 inhibitor GDC-0199 PO QD on days 1-28. GDC-0199 is administered through a dose ramp-up throughout course 3 with 20 mg administered in week 1, 50mg in week 2, 100mg in week 3 and 200mg in week 4. The 200mg dose level continues through the rest of the treatment period. Treatment repeats every 28 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.
  Bcl-2 Inhibitor GDC-0199: Given PO
  Obinutuzumab: Given IV
  Ibrutinib: Given PO
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
- Phase 1b Cohort 400mg Venetoclax (GDC-0199); Phase 2 Relapsed/Refractory; TN1: Phase 2 Treatment Naïve; TN2: Phase 2 Treatment Naïve: Patients receive obinutuzumab IV on day 1 (days 1, 2, 8, and 15 for course 1 only) every 28 days for up to 8 courses. Beginning in course 2, patients receive ibrutinib PO QD on days 1-28. Beginning in course 3, patients receive Bcl-2 inhibitor GDC-0199 PO QD on days 1-28. GDC-0199 is administered through a dose ramp-up throughout course 3 with 20 mg administered in week 1, 50mg in week 2, 100mg in week 3 and 200mg in week 4. The dose of GDC-0199 increases to 400mg starting week 1 of course 4. The 400mg dose level continues through the rest of the treatment period. Treatment repeats every 28 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.
  Bcl-2 Inhibitor GDC-0199: Given PO
  Obinutuzumab: Given IV
  Ibrutinib: Given PO
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
Period: Overall Study
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Started | 3 | 3 | 6 | 25 | 25 | 25
Completed | 3 | 3 | 6 | 22 | 21 | 24
Not Completed | 0 | 0 | 0 | 3 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve | Total
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 6 | 19 | 18 | 20 | 67
  >=65 years | 1 | 1 | 0 | 6 | 7 | 5 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 9 | 10 | 8 | 28
  Male | 3 | 3 | 5 | 16 | 15 | 17 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 6 | 25 | 24 | 23 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1 | 2
  White | 3 | 3 | 6 | 23 | 25 | 22 | 82
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 25 | 25 | 25 | 87

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Bcl-2 Inhibitor GDC-0199 in Combination With Obinutuzumab and Ibrutinib (Phase Ib)
Time Frame: 28 days (course 3)
Population: Maximum tolerated dose was only analyzed for phase l
Measure: Number; unit: milligrams
Groups:
- Phase 1b Cohort; Phase 2 Relapsed/Refractory; TN1: Phase 2 Treatment Naïve; TN2: Phase 2 Treatment Naïve: Patients receive obinutuzumab IV on day 1 (days 1, 2, 8, and 15 for course 1 only) every 28 days for up to 8 courses. Beginning in course 2, patients receive ibrutinib PO QD on days 1-28. Beginning in course 3, patients receive Bcl-2 inhibitor GDC-0199 PO QD on days 1-28. Treatment repeats every 28 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.
  Bcl-2 Inhibitor GDC-0199: Given PO
  Obinutuzumab: Given IV
  Ibrutinib: Given PO
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Phase 1b Cohort | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 12 | 0 | 0 | 0
milligrams | 400 |  |  |

2. Primary Outcome: Minimal Residual Disease (MRD)-Complete Response (CR) Defined by the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 Criteria (Phase II)
Description: Assessments of MRD will be used in patients classified as CR to further evaluate their status as disease-free and if this further impacts their ability to remain progression-free and alive. MRD will be determined by high sensitivity 4 color flow cytometric analysis of the bone marrow using validated panels.
Time Frame: Up to 8 weeks post-treatment
Population: MRD was only measured for phase 2 of the study
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b Cohort | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 0 | 25 | 25 | 25
percentage of participants |  | 44 | 56 | 60

3. Secondary Outcome: Number of Adverse Events Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: For all patients who receive at least one day of treatment, toxicities will be tabulated by type and grade and displayed in summary form. Serious adverse events are listed with "(SAE)" after the event name.
Time Frame: Up to 4 years
Measure: Number; unit: Number of Events
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
Number of Events
  Abdominal pain | 5 | 1 | 1 | 11 | 7 | 6
  Alanine Aminotransferase Increased | 2 | 4 | 8 | 23 | 12 | 23
  Alkaline Phosphatase Increased | 2 | 0 | 0 | 6 | 10 | 15
  Allergic Reaction | 1 | 0 | 0 | 0 | 5 | 2
  Allergic Rhinitis | 2 | 3 | 3 | 17 | 24 | 3
  Alopecia | 0 | 0 | 0 | 1 | 1 | 3
  Anemia | 4 | 0 | 0 | 20 | 28 | 16
  Anorexia | 0 | 2 | 2 | 10 | 21 | 14
  Anxiety | 0 | 1 | 3 | 14 | 9 | 2
  Arthralgia | 4 | 5 | 10 | 33 | 37 | 19
  Arthritis | 2 | 1 | 5 | 6 | 12 | 1
  Aspartate Aminotransferase Increased | 2 | 3 | 11 | 35 | 22 | 40
  Atrial Fibrillation | 0 | 0 | 0 | 2 | 4 | 5
  Back Pain | 3 | 3 | 1 | 16 | 22 | 13
  Blood Bilirubin Increased | 6 | 0 | 1 | 24 | 43 | 54
  Bloating | 1 | 0 | 0 | 1 | 1 | 8
  Blurred Vision | 0 | 0 | 4 | 8 | 11 | 3
  Bone Pain | 0 | 0 | 2 | 4 | 5 | 3
  Bronchial Infection | 1 | 4 | 0 | 7 | 3 | 2
  Bruising | 3 | 6 | 12 | 34 | 33 | 30
  Bullous Dermatitis | 2 | 1 | 0 | 1 | 3 | 1
  Cataract | 0 | 0 | 0 | 3 | 1 | 5
  Non-cardiac Chest Pain | 0 | 0 | 1 | 11 | 5 | 9
  Chest Pain - Cardiac | 0 | 0 | 1 | 4 | 2 | 1
  Chills | 1 | 1 | 0 | 14 | 20 | 10
  High Cholesterol | 1 | 0 | 1 | 7 | 4 | 1
  Chronic Kidney Disease | 2 | 0 | 1 | 4 | 0 | 1
  Confusion | 0 | 0 | 1 | 0 | 3 | 2
  Conjunctivitis | 1 | 0 | 0 | 2 | 2 | 2
  Constipation | 2 | 2 | 4 | 24 | 32 | 18
  Cough | 2 | 2 | 4 | 32 | 26 | 21
  Creatinine Increased | 7 | 7 | 8 | 32 | 27 | 25
  Dental Caries | 1 | 0 | 2 | 9 | 1 | 1
  Depression | 0 | 0 | 1 | 9 | 6 | 1
  Diarrhea | 4 | 5 | 16 | 46 | 44 | 63
  Dizziness | 2 | 1 | 6 | 11 | 19 | 16
  Dry Eyes | 1 | 0 | 1 | 5 | 4 | 6
  Dry Mouth | 1 | 0 | 2 | 1 | 3 | 1
  Dry Skin | 1 | 0 | 3 | 10 | 9 | 7
  Dysgeusia | 0 | 1 | 1 | 5 | 6 | 7
  Dyspepsia | 2 | 4 | 5 | 29 | 44 | 14
  Dysphagia | 0 | 0 | 0 | 3 | 3 | 1
  Dyspnea | 1 | 5 | 11 | 23 | 25 | 14
  Ear Pain | 0 | 0 | 0 | 2 | 5 | 4
  Epistaxis | 0 | 0 | 11 | 17 | 21 | 2
  Fall | 0 | 0 | 2 | 10 | 10 | 5
  Fatigue | 4 | 19 | 24 | 66 | 76 | 39
  Fever | 3 | 0 | 3 | 15 | 17 | 10
  Flatulence | 0 | 2 | 1 | 1 | 0 | 2
  Floaters | 0 | 0 | 1 | 2 | 0 | 2
  Flu Like Symptoms | 0 | 5 | 5 | 6 | 6 | 21
  Flushing | 0 | 0 | 1 | 1 | 2 | 2
  Gastroesophageal Reflux Disease | 0 | 1 | 4 | 2 | 1 | 3
  Headache | 5 | 6 | 6 | 35 | 27 | 23
  Hearing Impaired | 0 | 0 | 0 | 2 | 1 | 0
  Heamaturia | 1 | 0 | 0 | 5 | 8 | 3
  Hemorrhoids | 0 | 1 | 2 | 1 | 2 | 1
  Hot Flashes | 0 | 0 | 0 | 2 | 6 | 3
  Hyperglycemia | 5 | 0 | 7 | 53 | 40 | 31
  Hyperhidrosis | 4 | 7 | 4 | 17 | 24 | 12
  Hyperkalemia | 2 | 1 | 0 | 6 | 0 | 7
  Hypernatremia | 4 | 2 | 1 | 13 | 13 | 3
  Hypertension | 17 | 26 | 52 | 225 | 207 | 125
  Hyperuricemia | 6 | 5 | 20 | 55 | 37 | 28
  Hypoalbuminemia | 0 | 1 | 2 | 15 | 53 | 9
  Hypocalcemia | 3 | 17 | 11 | 74 | 98 | 56
  Hypoglycemia | 0 | 0 | 0 | 22 | 21 | 8
  Hypokalemia | 3 | 1 | 0 | 28 | 40 | 24
  Hypomagnesemia | 0 | 1 | 0 | 11 | 14 | 12
  Hyponatremia | 1 | 0 | 0 | 19 | 16 | 18
  Hypophosphatemia | 5 | 5 | 13 | 19 | 11 | 14
  Hypothyroidism | 0 | 0 | 1 | 1 | 3 | 1
  Infusion Related Reaction | 3 | 6 | 4 | 21 | 25 | 25
  Insomnia | 1 | 5 | 6 | 11 | 23 | 13
  Joint Range of Motion Decreased | 0 | 0 | 0 | 1 | 1 | 2
  Leukocytosis | 2 | 0 | 0 | 2 | 3 | 2
  Lung Infection | 0 | 2 | 2 | 4 | 5 | 8
  Lymph Node Pain | 1 | 1 | 0 | 3 | 5 | 1
  Lymphocyte Count Decreased | 24 | 29 | 30 | 170 | 162 | 172
  Lymphocyte Count Increased | 5 | 3 | 1 | 34 | 22 | 31
  Malaise | 0 | 0 | 0 | 1 | 5 | 4
  Mucositis Oral | 0 | 5 | 4 | 25 | 42 | 33
  Myalgia | 3 | 1 | 13 | 41 | 40 | 29
  Nail Loss | 0 | 2 | 1 | 8 | 6 | 0
  Nasal Congestion | 2 | 2 | 3 | 12 | 10 | 10
  Nausea | 1 | 2 | 8 | 32 | 41 | 34
  Neck Pain | 1 | 2 | 0 | 1 | 5 | 2
  Neutrophil Count Decreased | 18 | 34 | 24 | 229 | 169 | 169
  Oral Pain | 0 | 0 | 1 | 1 | 7 | 0
  Otitis Media | 0 | 0 | 0 | 3 | 3 | 5
  Pain | 4 | 0 | 6 | 9 | 8 | 6
  Palpitations | 0 | 0 | 0 | 7 | 4 | 7
  Paresthesia | 1 | 3 | 2 | 15 | 21 | 19
  Peripheral Sensory Neuropathy | 0 | 1 | 3 | 4 | 2 | 1
  Platelet Count Decreased | 21 | 12 | 58 | 177 | 175 | 103
  Postnasal Drip | 1 | 0 | 1 | 12 | 7 | 7
  Productive Cough | 0 | 0 | 0 | 6 | 1 | 6
  Proteinuria | 0 | 0 | 0 | 4 | 1 | 1
  Pruritus | 1 | 1 | 0 | 2 | 3 | 7
  Rash Acneiform | 0 | 0 | 0 | 3 | 5 | 3
  Rash Maculo-papular | 2 | 1 | 4 | 23 | 33 | 12
  Sinus Bradycardia | 1 | 0 | 2 | 36 | 20 | 29
  Sinus Disorder | 0 | 0 | 0 | 6 | 1 | 1
  Sinus Pain | 0 | 0 | 0 | 4 | 2 | 0
  Sinus Tachycardia | 1 | 0 | 0 | 9 | 5 | 10
  Sinusitis | 2 | 4 | 2 | 35 | 25 | 15
  Skin Infection | 1 | 0 | 8 | 13 | 11 | 6
  Sleep Apnea | 0 | 1 | 2 | 2 | 2 | 1
  Sore Throat | 0 | 1 | 3 | 12 | 17 | 11
  Syncope | 0 | 0 | 0 | 2 | 2 | 1
  Testicular Pain | 2 | 0 | 1 | 0 | 1 | 2
  Tinnitus | 0 | 0 | 0 | 7 | 4 | 2
  Toothache | 2 | 0 | 1 | 5 | 3 | 4
  Tremor | 0 | 0 | 1 | 0 | 1 | 4
  Upper Respiratory Infection | 5 | 5 | 8 | 30 | 28 | 11
  Urinary Frequency | 2 | 1 | 0 | 5 | 8 | 5
  Urinary Tract Infection | 0 | 0 | 2 | 6 | 20 | 3
  Vomiting | 0 | 2 | 3 | 19 | 10 | 12
  White Blood Cell Decreased | 19 | 34 | 24 | 231 | 184 | 186
  Weight Gain | 7 | 13 | 6 | 42 | 57 | 51
  Weight Loss | 1 | 2 | 10 | 11 | 10 | 8
  Activated partial thromboplastin time prolonged | 2 | 0 | 1 | 1 | 0 | 0
  Blood and lymphatic system disorders - Other | 1 | 1 | 0 | 2 | 0 | 3
  Ear and labyrinth disorders - Other | 1 | 0 | 0 | 6 | 2 | 5
  Eye Disorders - Other | 1 | 1 | 0 | 6 | 3 | 12
  Flank Pain | 1 | 0 | 0 | 0 | 1 | 2
  Gastrointestinal disorders - Other | 2 | 0 | 2 | 14 | 18 | 8
  Gum Infection | 2 | 0 | 0 | 0 | 0 | 2
  Injury, poisoning and procedural complications - Other | 1 | 1 | 11 | 9 | 17 | 10
  Musculoskeletal and connective tissue disorder - Other | 5 | 4 | 6 | 17 | 8 | 7
  Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other | 2 | 3 | 3 | 29 | 28 | 37
  Pain in Extremity | 1 | 1 | 2 | 22 | 13 | 9
  Pneumonitis | 2 | 0 | 0 | 0 | 3 | 0
  Renal and urinary disorders - Other | 2 | 0 | 0 | 1 | 1 | 0
  Skin and subcutaneous tissue disorders - Other | 4 | 2 | 12 | 24 | 23 | 29
  Surgical and medical procedures - Other | 1 | 0 | 0 | 0 | 1 | 0
  Urinary Retention | 1 | 0 | 0 | 3 | 0 | 2
  Vascular disorders - Other | 2 | 0 | 0 | 1 | 1 | 1
  Atrioventricular block complete | 0 | 1 | 0 | 0 | 0 | 0
  Cognitive Disturbance | 0 | 1 | 0 | 0 | 1 | 0
  Eye Infection | 0 | 1 | 0 | 0 | 1 | 0
  General disorders and administration site conditions - Other | 0 | 1 | 0 | 1 | 0 | 1
  Hypertriglyceridemia | 0 | 1 | 0 | 0 | 0 | 1
  Infections and infestations - Other | 0 | 1 | 3 | 17 | 28 | 35
  Memory Impairment | 0 | 1 | 0 | 0 | 1 | 0
  Metabolism and nutrition disorders - Other | 0 | 1 | 2 | 0 | 0 | 1
  Nail Ridging | 0 | 1 | 0 | 0 | 0 | 1
  Reproductive system and breast disorders - Other | 0 | 1 | 0 | 1 | 2 | 5
  Respiratory, thoracic and mediastinal disorders - Other | 0 | 2 | 0 | 1 | 2 | 0
  Rhinitis infective | 0 | 1 | 0 | 0 | 0 | 0
  Urinary Urgency | 0 | 1 | 0 | 0 | 0 | 1
  Anal Hemorrhage | 0 | 0 | 1 | 1 | 0 | 1
  Bladder Spasm | 0 | 0 | 1 | 0 | 1 | 0
  Cardiac Disorders - Other | 0 | 0 | 1 | 3 | 4 | 1
  Dysarthria | 0 | 0 | 3 | 0 | 1 | 0
  Edema Cerebral | 0 | 0 | 1 | 0 | 0 | 0
  Edema Face | 0 | 0 | 2 | 1 | 0 | 1
  Edema Limbs | 0 | 0 | 2 | 9 | 8 | 10
  Flashing Lights | 0 | 0 | 1 | 1 | 0 | 0
  Gastrointestinal Pain | 0 | 0 | 1 | 2 | 0 | 1
  Hematoma | 0 | 0 | 1 | 0 | 0 | 4
  Hypersomnia | 0 | 0 | 2 | 0 | 0 | 1
  Investigations - Other | 0 | 0 | 1 | 0 | 0 | 1
  Localized Edema | 0 | 0 | 1 | 18 | 15 | 8
  Osteoporosis | 0 | 0 | 1 | 0 | 1 | 2
  Periorbital Edema | 0 | 0 | 1 | 0 | 0 | 0
  Rectal Hemorrhage | 0 | 0 | 1 | 1 | 0 | 0
  Stomach Pain | 0 | 0 | 1 | 1 | 1 | 0
  Tooth Infection | 0 | 0 | 1 | 0 | 1 | 1
  Urinary Tract Pain | 0 | 0 | 2 | 0 | 0 | 0
  Vaginal Infection | 0 | 0 | 1 | 0 | 2 | 0
  Vertigo | 0 | 0 | 1 | 0 | 0 | 2
  Cholecystitis | 0 | 0 | 0 | 3 | 0 | 0
  Laryngeal inflammation | 0 | 0 | 0 | 4 | 0 | 1
  Nail Infection | 0 | 0 | 0 | 3 | 3 | 0
  Oral Hemorrhage | 0 | 0 | 0 | 2 | 2 | 0
  Otitis Externa | 0 | 0 | 0 | 2 | 1 | 1
  Purpura | 0 | 0 | 0 | 3 | 3 | 1
  Watering Eyes | 0 | 0 | 0 | 2 | 0 | 0
  Fracture | 0 | 0 | 0 | 1 | 3 | 0
  Generalized Muscle Weakness | 0 | 0 | 0 | 0 | 4 | 0
  Hoarseness | 0 | 0 | 0 | 0 | 3 | 2
  Muscle Weakness Lower Limb | 0 | 0 | 0 | 1 | 3 | 0
  Agitation | 0 | 0 | 0 | 0 | 1 | 2
  Chest Wall Pain | 0 | 0 | 0 | 1 | 0 | 2
  Erectile Dysfunction | 0 | 0 | 0 | 1 | 0 | 2
  Hiccups | 0 | 0 | 0 | 1 | 0 | 2
  INR increased | 0 | 0 | 0 | 0 | 0 | 2
  Nervous system disorders - Other | 0 | 0 | 0 | 2 | 1 | 2
  Neuralgia | 0 | 0 | 0 | 0 | 1 | 2
  Paronychia | 0 | 0 | 0 | 5 | 2 | 2
  Blood and lymphatic system disorders - other (SAE) | 0 | 0 | 0 | 0 | 0 | 1
  Febrile neutropenia | 0 | 0 | 0 | 1 | 0 | 1
  Atrial fibrillation (SAE) | 0 | 0 | 0 | 0 | 2 | 1
  Atrioventricular block complete (SAE) | 0 | 1 | 0 | 0 | 0 | 0
  Cardiac disorders - Other (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Chest pain - cardiac (SAE) | 0 | 0 | 0 | 2 | 0 | 0
  Abdominal pain (SAE) | 1 | 0 | 0 | 0 | 0 | 0
  Colitis (SAE) | 0 | 0 | 0 | 0 | 1 | 0
  Fatigue (SAE) | 0 | 0 | 0 | 1 | 1 | 0
  Fever (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Flu like symptoms (SAE) | 0 | 1 | 0 | 0 | 0 | 0
  Cholecystitis (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Bronchial infection (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Infections and infestations - other (SAE) | 0 | 1 | 1 | 0 | 0 | 3
  Lung Infection (SAE) | 0 | 1 | 1 | 1 | 1 | 2
  Sepsis (SAE) | 0 | 0 | 0 | 0 | 1 | 0
  Sinusitis (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Skin infection (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Upper Respiratory Infection (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Infusion related reaction (SAE) | 0 | 0 | 0 | 0 | 0 | 1
  Stroke (SAE) | 0 | 0 | 0 | 0 | 0 | 1
  Alanine Aminotransferase increased (SAE) | 0 | 0 | 0 | 0 | 1 | 0
  Aspartate aminotransferase increased (SAE) | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophil count decreased (SAE) | 0 | 0 | 0 | 0 | 0 | 4
  Dehydration (SAE) | 0 | 0 | 0 | 0 | 1 | 0
  Hyperkalemia (SAE) | 0 | 0 | 0 | 0 | 0 | 2
  Hypoglycemia (SAE) | 0 | 0 | 0 | 0 | 1 | 0
  Metabolism and nutrition disorders - other (SAE) | 0 | 0 | 0 | 0 | 0 | 1
  Tumor lysis syndrome (SAE) | 0 | 0 | 0 | 0 | 0 | 1
  Pain in extremity (SAE) | 0 | 0 | 0 | 1 | 1 | 0
  Headache (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Nervous system disorders - other (SAE) | 0 | 0 | 0 | 1 | 1 | 0
  Syncope (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Pneumonitis (SAE) | 0 | 0 | 0 | 0 | 1 | 0
  Wheezing (SAE) | 0 | 0 | 0 | 1 | 0 | 0
  Hyperhidrosis (SAE) | 0 | 0 | 0 | 0 | 0 | 1
  Hypertension (SAE) | 0 | 1 | 0 | 1 | 0 | 0

4. Secondary Outcome: Number of Courses Started/Completed
Description: May be summarized.
Time Frame: Up to 14 months
Measure: Number; unit: number of subjects
Groups:
- Phase 1b Cohort 100mg Venetoclax (GDC-0199): Patients receive obinutuzumab IV on day 1 (days 1, 2, 8, and 15 for course 1 only) every 28 days for up to 8 courses. Beginning in course 2, patients receive ibrutinib PO QD on days 1-28. Beginning in course 3, patients receive Bcl-2 inhibitor GDC-0199 PO QD on days 1-28. GDC-0199 is administered through a dose ramp-up throughout course 3 with 20 mg administered in week 1, 50mg in week 2 and 100mg in week 3. The 100mg dose level continues through the rest of the treatment period. Treatment repeats every 28 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.
  Bcl-2 Inhibitor GDC-0199: Given PO Obinutuzumab: Given IV Ibrutinib: Given PO Pharmacological Study: Correlative studies Laboratory Biomarker Analysis: Correlative studies Quality-of-Life Assessment: Ancillary studies
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
number of subjects
  Completed 14 cycles | 3 | 3 | 6 | 22 | 21 | 24
  Completed 13 or less cycles | 0 | 0 | 0 | 3 | 4 | 1

5. Secondary Outcome: Number of Patients Who Reach the Target Dose of Bcl-2 Inhibitor GDC-0199
Description: May be summarized.
Time Frame: Up to 14 months
Population: Target dose of Bcl-2 inhibitor GDC-0199 only measured for Phase ll subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 0 | 25 | 25 | 25
Participants |  | 24 | 25 | 25

6. Secondary Outcome: Number of Patients Requiring Dose Reductions
Description: May be summarized.
Time Frame: Up to 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
Participants | 0 | 0 | 0 | 2 | 0 | 5

7. Secondary Outcome: Reason for Going Off Treatment
Description: May be summarized.
Time Frame: Up to 14 months
Measure: Number; unit: participants
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
participants
  Adverse Event | 0 | 0 | 0 | 1 | 2 | 1
  Physician Decision | 0 | 0 | 0 | 2 | 2 | 0
  Treatment completed per protocol | 3 | 3 | 6 | 22 | 21 | 24

8. Secondary Outcome: Overall Response Rate
Description: Overall response rate will be reported for all evaluable patients in the phase II setting, within and potentially across cohorts, assuming a binomial distribution.
Time Frame: Up to 4 years
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
percentage of participants | 66.7 | 100 | 100 | 88 | 84 | 96

9. Secondary Outcome: Progression-free Survival (PFS)
Description: Will be summarized by the Kaplan-Meier method for each of the phase II cohorts.
Time Frame: Time from first treatment date until the date of progression or death, whichever occurs first, assessed up to 8 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
months | NA [NA to NA] — For the phase 1b cohort, median PFS was not reached due to an insufficient number of events | NA [NA to NA] — For the phase 1b cohort, median PFS was not reached due to an insufficient number of events | NA [NA to NA] — For the phase 1b cohort, median PFS was not reached due to an insufficient number of events | 81.8 [57.3 to NA] — The upper limit of the confidence interval was not reached due to not enough participants experiencing progression or death | 88.5 [80.6 to NA] — The upper limit of the confidence interval was not reached due to not enough participants experiencing progression or death | NA [NA to NA] — For the TN2 cohort, median PFS was not reached due to an insufficient number of events

10. Secondary Outcome: Emotional Distress Assessment
Description: Validated instruments will be administered serially to assess longitudinal changes in measures of health related quality of life using 36-Item Short Form Survey (SF-36) Mental Component Scale (MCS) T-scores for each time point with pairwise comparison p-values. Scores on the SF-36 scale range from 0 to 100, with higher scores indicating better mental health. Scores for the MCS are standardized using U.S. general population norms with summary scores set relative to a t-score mean of 50 and a standard deviation of 10.
Time Frame: Cycle 1 day 1, cycle 2 day 1, cycle 3 day 1, cycle 6 day 1 and cycle 12 day 1
Population: In the phase 1b study, as not all patients were treated at the target dose of venetoclax, psychologic outcomes were not planned to be collected. In the newest cohort (the TN2 cohort) these studies were similarly not planned or included as adequate information had been gained on the outcomes measures from the original phase 2 cohorts.
  The number of analyzed participants at each time point represents the number of participants who completed the survey at that time point.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 0 | 0 | 0 | 21 | 23 | 0
T-score
  Cycle 1 Day 1 |  |  |  | 54.03 (9.25) | 52.32 (6.87) |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 20 | 21 | 0
  Cycle 2 Day 1 |  |  |  | 54.42 (7.75) | 54.88 (6.10) |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 20 | 21 | 0
  Cycle 3 Day 1 |  |  |  | 55.90 (7.05) | 54.33 (6.54) |
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 18 | 23 | 0
  Cycle 6 Day 1 |  |  |  | 56.31 (7.64) | 53.50 (8.96) |
  Cycle 12 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 14 | 17 | 0
  Cycle 12 Day 1 |  |  |  | 55.53 (5.34) | 54.35 (6.30) |

11. Secondary Outcome: Health Related Quality of Life
Description: Validated instruments will be administered serially to assess longitudinal changes in measures of health related quality of life using 36-Item Short Form Survey (SF-36) Physical Component Scale (PCS) T-scores for each time point with pairwise comparison p-values. Scores on the SF-36 scale range from 0 to 100, with higher scores indicating better physical health. Scores for the PCS are standardized using U.S. general population norms with summary scores set relative to a t-score mean of 50 and a standard deviation of 10.
Time Frame: Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 6 Day 1, and Cycle 12 Day 1 (each cycle is 28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 1b Cohort | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 0 | 21 | 23 | 0
T-score
  Cycle 1 Day 1 |  | 42.88 (12.52) | 44.25 (10.97) |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 20 | 21 | 0
  Cycle 2 Day 1 |  | 45.53 (12.12) | 42.01 (10.57) |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 20 | 21 | 0
  Cycle 3 Day 1 |  | 45.17 (13.56) | 44.92 (11.86) |
  Cycle 6 Day 1: number analyzed (Participants) | 0 | 18 | 23 | 0
  Cycle 6 Day 1 |  | 45.94 (12.95) | 46.75 (11.37) |
  Cycle 12 Day 1: number analyzed (Participants) | 0 | 14 | 17 | 0
  Cycle 12 Day 1 |  | 45.97 (14.05) | 46.40 (11.45) |

12. Secondary Outcome: Serial Assessment of Immune Effector Cell Number and Function.
Description: Peripheral blood immunophenotyping will be used to enumerate immune effector cells (counts and percentages of T-, and Natural Killer (NK)-cell subsets).
Time Frame: 4 weeks post-treatment
Population: In the phase 1b study, as not all patients were treated at the target dose of venetoclax, immune cell subsets were not planned to be collected. In the TN2 cohort these studies were similarly not planned or included as adequate information had been gained on the outcomes measures from the original phase 2 cohorts. Five participants from the Phase 2 RR cohort and four participants from the TN1 cohort did not complete treatment or were unable to have data collected for immune cell subsets.
Measure: Mean (Standard Deviation); unit: 10^3 cells/uL
Groups:
- Phase 2 Relapsed/Refractory (RR); TN1: Phase 2 Treatment Naïve; TN2: Phase 2 Treatment Naïve: Patients receive obinutuzumab IV on day 1 (days 1, 2, 8, and 15 for course 1 only) every 28 days for up to 8 courses. Beginning in course 2, patients receive ibrutinib PO QD on days 1-28. Beginning in course 3, patients receive Bcl-2 inhibitor GDC-0199 PO QD on days 1-28. Treatment repeats every 28 days for up to 14 courses in the absence of disease progression or unacceptable toxicity.
  Bcl-2 Inhibitor GDC-0199: Given PO
  Obinutuzumab: Given IV
  Ibrutinib: Given PO
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
Arm/Group | Phase 1b Cohort | Phase 2 Relapsed/Refractory (RR) | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 0 | 20 | 21 | 0
10^3 cells/uL
  NK |  | 95 (64) | 89 (49) |
  CD3+CD4+ |  | 499 (217) | 738 (298) |
  CD3+CD8+ |  | 479 (296) | 312 (213) |

13. Secondary Outcome: Baseline Prognostic Factors: Number of Prior Therapies
Description: Relationships between baseline prognostic factors and response may be screened and analyzed quantitatively using logistic regression and adjusting for disease cohort, particularly if a sufficient number of patients respond to this combination therapy.
Time Frame: Baseline
Measure: Median (Full Range); unit: Number of Prior Therapies
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
Number of Prior Therapies | 1 [1 to 7] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 3] | 0 [0 to 0] | 0 [0 to 0]

14. Secondary Outcome: Baseline Prognostic Factors: Tumor Lysis Syndrome (TLS) Risk
Description: as for outcome 13
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
participants
  TLS Risk Low | 0 | 0 | 1 | 7 | 1 | 1
  TLS Risk Medium | 2 | 3 | 2 | 8 | 18 | 17
  TLS Risk High | 1 | 0 | 3 | 10 | 6 | 7

15. Secondary Outcome: Baseline Prognostic Factors: Hemoglobin
Time Frame: Baseline
Population: One participant in the TN2 cohort did not have hemoglobin measured at baseline.
Measure: Median (Full Range); unit: grams per deciliter
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 24
grams per deciliter | 12.3 [12.3 to 13.3] | 11.4 [11.2 to 12.7] | 12.7 [11.6 to 15.8] | 12 [9 to 16] | 10 [8 to 13] | 10 [7 to 15]

16. Secondary Outcome: Baseline Prognostic Factors: Investigations
Description: Absolute neutrophil count (ANC), Absolute lymphocyte count (ALC) and Platelets.
Time Frame: Baseline
Measure: Median (Full Range); unit: 10^3 cells/uL
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
10^3 cells/uL
  Platelets | 117 [103 to 227] | 158 [102 to 208] | 171.5 [139 to 222] | 132 [52 to 255] | 166 [68 to 231] | 132 [23 to 488]
  ANC | 8.9 [0.2 to 23.5] | 2.6 [0 to 5.1] | 5.5 [3.2 to 9.9] | 3 [1 to 28] | 5 [1 to 26] | 4 [1 to 16]
  ALC | 135.3 [19.6 to 445.6] | 144.9 [79.2 to 230.6] | 30.0 [2.8 to 287.2] | 29 [0 to 348] | 109 [3 to 413] | 191 [3 to 488]

17. Secondary Outcome: Baseline Prognostic Factor: Beta-2-microglobulin (B2M)
Description: Beta-2-microglobulin (B2M)
Time Frame: At baseline
Measure: Median (Full Range); unit: milligrams per liter
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
milligrams per liter | 5.2 [3.9 to 6.8] | 4.2 [2.7 to 5.0] | 2.6 [2.2 to 3.4] | 4 [2 to 7] | 3 [2 to 7] | 3 [2 to 6]

18. Secondary Outcome: Baseline Prognostic Factors: Lactate Dehydrogenase (LDH)
Description: lactate dehydrogenase (LDH)
Time Frame: At baseline
Measure: Median (Full Range); unit: units per liter
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
units per liter | 293 [219 to 371] | 301 [237 to 410] | 202 [155 to 899] | 223 [131 to 725] | 230 [98 to 710] | 280 [147 to 921]

19. Secondary Outcome: Baseline Prognostic Factors: Genetic Factors
Time Frame: At baseline
Population: The number of participants analyzed for each genetic factor represents the number of participants for which data was available for that genetic factor. The number of participants with High Hyperdiploid (HeH), was not a prespecified baseline measure so data was not collected for the phase 1b cohorts.
Measure: Number; unit: participants
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
Number analyzed (Participants) | 3 | 3 | 6 | 25 | 25 | 25
participants
  High Hyperdiploid (HeH): number analyzed (Participants) | 0 | 0 | 0 | 24 | 24 | 25
  High Hyperdiploid (HeH) |  |  |  | 19 | 17 | 19
  Zap-70 methylated: number analyzed (Participants) | 3 | 3 | 6 | 22 | 22 | 10
  Zap-70 methylated | 0 | 1 | 4 | 11 | 8 | 3
  Complex karyotype: number analyzed (Participants) | 3 | 3 | 6 | 24 | 25 | 25
  Complex karyotype | 1 | 1 | 3 | 8 | 8 | 11
  del(17p) | 0 | 0 | 1 | 1 | 3 | 2
  del(11q) | 3 | 1 | 4 | 9 | 5 | 7
  trisomy 12 | 0 | 0 | 1 | 4 | 3 | 3
  del(13q) | 2 | 0 | 2 | 0 | 5 | 16

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: All treatment arms were combined for adverse event reporting, since all arms received the same treatment regimen.
Arm/Group | Phase 1b Cohort 100mg Venetoclax (GDC-0199) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) | Phase 2 Relapsed/Refractory | TN1: Phase 2 Treatment Naïve | TN2: Phase 2 Treatment Naïve
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/3 | 0/6 | 1/25 | 1/25 | 1/25
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 2/6 | 12/25 | 7/25 | 11/25
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 25/25 | 25/25 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Cohort 100mg Venetoclax (GDC-0199) (N=3) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) (N=3) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) (N=6) | Phase 2 Relapsed/Refractory (N=25) | TN1: Phase 2 Treatment Naïve (N=25) | TN2: Phase 2 Treatment Naïve (N=25)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 3 (3)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (4)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Stroke (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1b Cohort 100mg Venetoclax (GDC-0199) (N=3) | Phase 1b Cohort 200mg Venetoclax (GDC-0199) (N=3) | Phase 1b Cohort 400mg Venetoclax (GDC-0199) (N=6) | Phase 2 Relapsed/Refractory (N=25) | TN1: Phase 2 Treatment Naïve (N=25) | TN2: Phase 2 Treatment Naïve (N=25)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 1 (1) | 1 (1) | 7 (11) | 6 (7) | 4 (6)
Alanine Aminotransferase increased (Investigations) | 2 (2) | 3 (4) | 4 (8) | 10 (23) | 8 (12) | 13 (23)
Alkaline Phosphatase Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 3 (6) | 6 (10) | 7 (15)
Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3) | 3 (3) | 13 (17) | 15 (24) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0) | 0 (0) | 12 (20) | 10 (28) | 5 (16)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (2) | 10 (10) | 14 (21) | 12 (14)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3) | 11 (14) | 8 (9) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (5) | 5 (10) | 13 (33) | 17 (37) | 9 (19)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (5) | 5 (6) | 10 (12) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 2 (2) | 3 (3) | 3 (11) | 13 (35) | 12 (22) | 17 (40)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 3 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (3) | 1 (1) | 10 (16) | 14 (22) | 6 (13)
Blood Bilirubin Increased (Investigations) | 2 (6) | 0 (0) | 1 (1) | 8 (24) | 12 (43) | 12 (54)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (8)
Blurred Vision (Eye disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (8) | 10 (11) | 3 (3)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 4 (5) | 3 (3)
Bronchial Infection (Infections and infestations) | 1 (1) | 2 (4) | 0 (0) | 5 (7) | 3 (3) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 3 (3) | 3 (6) | 6 (12) | 20 (34) | 19 (33) | 19 (30)
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (5)
Non-cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 8 (11) | 5 (5) | 5 (9)
Chest pain - Cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 10 (14) | 13 (20) | 9 (10)
High Cholesterol (Investigations) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 4 (4) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (2) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (2) | 2 (2) | 3 (4) | 12 (24) | 16 (32) | 8 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (4) | 13 (32) | 16 (26) | 13 (21)
Creatinine Increased (Investigations) | 2 (7) | 2 (7) | 1 (8) | 11 (32) | 9 (27) | 12 (25)
Dental Caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 7 (9) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (9) | 6 (6) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4) | 2 (5) | 6 (16) | 19 (46) | 17 (44) | 24 (63)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 5 (6) | 8 (11) | 12 (19) | 12 (16)
Dry Eyes (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (5) | 4 (4) | 6 (6)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 8 (10) | 8 (9) | 7 (7)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 2 (6) | 6 (7)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 2 (4) | 4 (5) | 16 (29) | 21 (44) | 8 (14)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (5) | 4 (11) | 15 (23) | 17 (25) | 9 (14)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (11) | 9 (17) | 11 (21) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 7 (10) | 8 (10) | 3 (5)
Fatigue (General disorders) | 3 (4) | 2 (19) | 6 (24) | 21 (66) | 23 (76) | 17 (39)
Fever (General disorders) | 2 (3) | 0 (0) | 2 (3) | 10 (15) | 6 (17) | 7 (10)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Flu like Symptoms (General disorders) | 0 (0) | 2 (5) | 4 (5) | 6 (6) | 4 (6) | 11 (21)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 2 (5) | 2 (6) | 5 (6) | 14 (35) | 16 (27) | 15 (23)
Hearing Impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 7 (8) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 1 (1)
Hot Flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 6 (6) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 5 (7) | 16 (53) | 18 (40) | 14 (31)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (7) | 2 (4) | 10 (17) | 12 (24) | 7 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0) | 3 (6) | 0 (0) | 5 (7)
Hypernatremia (Metabolism and nutrition disorders) | 1 (4) | 2 (2) | 1 (1) | 9 (13) | 6 (13) | 3 (3)
Hypertension (Vascular disorders) | 3 (17) | 3 (26) | 6 (52) | 25 (225) | 25 (207) | 22 (125)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (6) | 2 (5) | 5 (20) | 18 (55) | 15 (37) | 12 (28)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 8 (15) | 13 (53) | 4 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 3 (17) | 5 (11) | 21 (74) | 20 (98) | 18 (56)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (22) | 7 (21) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 10 (28) | 12 (40) | 10 (24)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (11) | 5 (14) | 6 (12)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (19) | 6 (16) | 5 (18)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (5) | 2 (5) | 4 (13) | 7 (19) | 6 (11) | 6 (14)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 3 (3) | 3 (6) | 4 (4) | 17 (21) | 20 (25) | 21 (25)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (5) | 4 (6) | 8 (11) | 16 (23) | 10 (13)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Lung Infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 2 (4) | 4 (5) | 4 (8)
Lymph Node Pain (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 3 (24) | 3 (29) | 5 (30) | 23 (170) | 22 (162) | 25 (172)
Lymphocyte Count Increased (Investigations) | 2 (5) | 3 (3) | 1 (1) | 13 (34) | 15 (22) | 17 (31)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 4 (4)
Mucositis Oral (Gastrointestinal disorders) | 0 (0) | 2 (5) | 2 (4) | 13 (25) | 20 (42) | 15 (33)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 6 (13) | 19 (41) | 18 (40) | 15 (29)
Nail Loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 7 (8) | 6 (6) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) | 9 (12) | 6 (10) | 7 (10)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (8) | 13 (32) | 18 (41) | 17 (34)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 4 (5) | 2 (2)
Neutrophil Count Decreased (Investigations) | 3 (18) | 3 (34) | 6 (24) | 24 (229) | 23 (169) | 24 (169)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (7) | 0 (0)
Otitis Media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 4 (5)
Pain (General disorders) | 2 (4) | 0 (0) | 3 (6) | 8 (9) | 6 (8) | 4 (6)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 4 (4) | 6 (7)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (3) | 2 (2) | 10 (15) | 13 (21) | 11 (19)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (21) | 3 (12) | 5 (58) | 22 (177) | 24 (175) | 22 (103)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 7 (12) | 6 (7) | 6 (7)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 4 (6)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 5 (7)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 4 (5) | 2 (3)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 2 (4) | 9 (23) | 18 (33) | 8 (12)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 13 (36) | 11 (20) | 11 (29)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 1 (1)
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (9) | 4 (5) | 6 (10)
Sinusitis (Infections and infestations) | 2 (2) | 2 (4) | 2 (2) | 15 (35) | 11 (25) | 9 (15)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (8) | 5 (13) | 5 (11) | 3 (6)
Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (3) | 9 (12) | 12 (17) | 8 (11)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Testicular Pain (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 3 (4) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 3 (5) | 3 (3) | 4 (4)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Upper Respiratory Infection (Infections and infestations) | 2 (5) | 3 (5) | 4 (8) | 12 (30) | 15 (28) | 8 (11)
Urinary Frequency (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 5 (5) | 8 (8) | 3 (5)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 3 (6) | 10 (20) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (3) | 9 (19) | 8 (10) | 8 (12)
White Blood Cell Decreased (Investigations) | 3 (19) | 3 (34) | 5 (24) | 24 (231) | 23 (184) | 24 (186)
Weight Gain (Investigations) | 3 (7) | 3 (13) | 3 (6) | 17 (42) | 20 (57) | 18 (51)
Weight Loss (Investigations) | 1 (1) | 1 (2) | 3 (10) | 8 (11) | 6 (10) | 7 (8)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 2 (2) | 4 (5)
Eye disorders - Other (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (6) | 3 (3) | 8 (12)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 11 (14) | 9 (18) | 7 (8)
Gum infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 5 (11) | 6 (9) | 10 (17) | 8 (10)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (4) | 3 (6) | 7 (17) | 6 (8) | 5 (7)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (3) | 3 (3) | 15 (29) | 11 (28) | 16 (37)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 10 (22) | 9 (13) | 7 (9)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2) | 5 (12) | 10 (24) | 14 (23) | 12 (29)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2)
Vascular disorders - Other (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 11 (17) | 12 (28) | 16 (35)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 4 (5)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4) | 1 (1)
Dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Edema cerebral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (9) | 8 (8) | 6 (10)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Hypersomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Investigations - Other (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 12 (18) | 10 (15) | 8 (8)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Periorbital edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Paronychia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT02427451/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02427451/ICF_001.pdf